CLINICAL TRIAL: NCT00339274
Title: The Chernobyl Tissue Bank
Brief Title: International Cooperation for Post-Cherynobyl NIS Thyroid Tissue and Data Banks
Status: Completed | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999900024; OH00-C-N024; NCT00897572 (obsolete NCT alias)
Record Dates: First submitted 2006-06-19; First posted 2006-06-21 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2012-03-16

CONDITIONS: Environment
Keywords: Repositories; Pathology; Belarus; Russia; Ukraine

SUMMARY:
The large number of thyroid tumors that have occurred in areas exposed to high levels of fallout from the Chernobyl accident raise problems of public health importance, or regulatory importance, and of scientific importance. The over-riding priority must go to matters such as diagnosis, treatment of those affected and prevention, and International Agencies are giving financial and material help in these areas. However providing the needs of the patient are not compromised, it is very important to ensure that information that may be of value to the health of future generations is not lost. International agencies are again providing financial support for a variety of joint studies, some of which are based on studies of tissues from thyroid operations carried out as part of treatment, and not required for the initial diagnosis on which treatment is based. An international coordinated approach to this problem is not in place to help Belarus, the Russian Federation and Ukraine to establish their own comprehensive thyroid tissue and data banks and to ensure that tissue and nucleic acids are used to contribute to the understanding of the consequences of the Chernobyl accident. This project has the support of the Governments of Belarus, the Russian Federation and Ukraine and the National Cancer Institute of the USA, (NCI), the European Commission (EC), the Sasakawa Memorial Health Foundation of Japan (SMHF) and the World Health Organization (WHO) have agreed to cooperate in supporting this project.

DETAILED DESCRIPTION:
The large number of thyroid tumors that have occurred in areas exposed to high levels of fallout from the Chernobyl accident raise problems of public health importance, or regulatory importance, and of scientific importance. The over-riding priority must go to matters such as diagnosis, treatment of those affected and prevention, and International Agencies are giving financial and material help in these areas. However providing the needs of the patient are not compromised, it is very important to ensure that information that may be of value to the health of future generations is not lost. International agencies are again providing financial support for a variety of joint studies, some of which are based on studies of tissues from thyroid operations carried out as part of treatment, and not required for the initial diagnosis on which treatment is based. An international coordinated approach to this problem is not in place to help Belarus, the Russian Federation and Ukraine to establish their own comprehensive thyroid tissue and data banks and to ensure that tissue and nucleic acids are used to contribute to the understanding of the consequences of the Chernobyl accident. This project has the support of the Governments of Belarus, the Russian Federation and Ukraine and the National Cancer Institute of the USA, (NCI), the European Commission (EC), the Sasakawa Memorial Health Foundation of Japan (SMHF) and the World Health Organization (WHO) have agreed to cooperate in supporting this project.

ELIGIBILITY:
* INCLUSION CRITERIA:

Patients with thyroid tumours from the whole of Belarus, and the contaminated oblasts of the Russian Federation and Ukraine who were born after 26th April 1967.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 4000 (Estimated)
Dates: Start 1999-10-14; Study Completion 2012-03-16

CONTACTS AND LOCATIONS:
Overall Officials: Louise Brinton, Ph.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Cancer Institute (NCI), 9000 Rockville Pike, Bethesda, Maryland, United States